CLINICAL TRIAL: NCT05088122
Title: Hormonal Effect Of Different Phases Of Menstrual Cycle On Postural Stability In Postpubertal Females: A Cross Sectional Repeated Measure Design
Brief Title: Hormonal Effect of Different Menstrual Phases on Dynamic Balance in Postpubertal Females
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hager Mohey Eldien Abdel Aziz Mahmoud, Demonstrator of physical therapy for women health at deraya university, Cairo University
Other Study IDs: P.T.REC/012/003102
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Menstrual Cycle
Keywords: Sex hormones, Postural stability, Menstrual cycle.

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention, not applicable

SUMMARY:
High rate of injuries detected during certain periods of menstrual cycle, raised the suggestion of the effecacy of the female sex hormones on soft tissue and neuromuscular control with subsequent deterioration of postural stability and high injury prevalence in post pubertal females so the aim of the present study is to investigate the effect of female sex hormones on postural stability in post pubertal females.

DETAILED DESCRIPTION:
Thirty-six post pubertal females will participate in this study. They will be selected from students and graduates of Faculty of Physical Therapy, Deraya University and they will be assigned into one group. Postural stability assessment will be carried out throughout three menstrual cycle phases, early follicular, ovulation and mid luteal phases by Biodex balance system. The timing of menstrual cycle phases will be determined by measuring serum estradiol and progesterone level. The exact time of ovulation will be determined by urine lutenizing hormone ovulatory strip test.

ELIGIBILITY:
Inclusion Criteria:

1. All females will be virginal.
2. Their ages will range from 15-25 years.
3. Their body mass index (BMI) will range from 18-27 kg/m2.
4. All females will have regular menstrual cycle within average of 28 days.

Exclusion Criteria:

1. Females having menstrual irregularity.
2. Use of oral contraceptives or any hormonal treatment in the previous six months before participate in this study.
3. History of lower extremity injury, surgery or pain during ADL.
4. Females having any vestibular problems , otitis media, labyrinthitis or any inner ear problems that affect balance.

Ages: 16 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Thirty-six, healthy postpubertal females , their ages will be ranged from 16-25 and BMI will be ranged from 18-27kg/m2, with regular menstrual cycle and with no any health condition that can affect the balance performance
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2021-12-25 (Estimated); Study Completion 2022-01-25 (Estimated)

PRIMARY OUTCOMES:
serum estradiol level | two months
  used for accurate timing of menstrual cycle phases, follicular and midluteal.
Anetro-posterior stability index | two months
  Indicator for dynamic postural stability
Medio-lateral stability index | two months
  Indicator for dynamic postural stability
Overall stability index | two months
  Indicator for dynamic postural stability

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF